CLINICAL TRIAL: NCT02125825
Title: Kinesia-D Phase II In-Clinic Continuous Assessment Study
Brief Title: Ambulatory Parkinson's Disease Dyskinesia Monitor for Drug Therapy Titration
Acronym: Kinesia-D
Status: Completed | Type: Observational
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); University of Rochester (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: KinesiaDPhaseIIYear1; 9R44AG044293 (NIH)
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Parkinson's disease on levodopa: Individuals with Parkinson's disease who are taking levodopa to treat motor symptoms

SUMMARY:
The objective is to assess a compact, portable, wireless movement disorder system with continuous monitoring capabilities to detect and quantify the severity of levodopa-induced dyskinesia in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease
* Clinical history of levodopa-induced dyskinesia
* 21 Years of age or older
* Stage 2 - 4 OFF-medication on the Hoehn and Yahr scale

Exclusion Criteria:

* Dementia (determined by a neuropsychological assessment)
* Severe tremor unaffected by levodopa

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Parkinson's disease and a history of levodopa-induced dyskinesia
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Correlation between motion sensor features and clinician-rated dyskinesia severity | All data will be collected within a single session not to exceed 3 hours
  Motor function (movement speed and magnitude measured with a motion sensor) will be collected for a period of 2 hours after taking normally prescribed dose of levodopa.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - University of Rochester Medical Center, Rochester, New York